CLINICAL TRIAL: NCT03241680
Title: Study of Anal Cytologies in Patients With High Grade Cervical Intraepithelial Neoplasia (CIN II and III)
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Universidade do Vale do Sapucai (Other)
Responsible Party: Principal Investigator, Lyliana Coutinho Resende Barbosa, MD Phd, Universidade do Vale do Sapucai
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: Citologia anal
Record Dates: First submitted 2017-08-02; First posted 2017-08-07 (Actual); Last update posted 2017-08-07 (Actual); Status verified 2017-08

CONDITIONS: Anal Carcinoma; Anal Condyloma
MeSH Terms: conditions — Anus Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Control Group with conventional citology (No Intervention): Patients who do not have high grade cervical intraepithelial neoplasia and will have anal cytology performed by conventional method
- Control Group with liquid based citology (No Intervention): Patients who do not have cervical intraepithelial neoplasia of high grade and will have anal cytology performed by liquid based method
- CIN 2-3/Conventional Citology (No Intervention): Patients with high grade cervical intraepithelial neoplasia and will have anal citology performed by conventional method
- CIN 2-3/Liquid Based (Active Comparator): Patients with high grade cervical intraepithelial neoplasia and will have anal citology performed by liquid based method
  Interventions: Diagnostic Test: Search of anal citology alterations

INTERVENTIONS:
Diagnostic Test: Search of anal citology alterations — All patients with a pathological diagnosis of CIN II and III, and in the general gynecological surgery outpatient clinic, will be selected at the outpatient clinic of Oncology Gynecology of the HCSL for a period of six months.
  Patients who meet the eligibility criteria will be clarified about the study, and only those who agree to participate will be included, by signing the informed consent form (TCLE).
  Arms: CIN 2-3/Liquid Based

SUMMARY:
Cervical cancer is the third most frequent neoplasm in Brazilian women (estimated risk of 15.33 cases / 100,000 women by 2014), behind breast and colorectal cancer.

This high incidence is explained by the pre-neoplastic lesions of the cervix being probably related to the practice of unsafe sex and to a poor local immune response against HPV.

Human papillomavirus (HPV) infection affects people of any age, although it is more common in young people, probably due to increased sexual activity in that period.

The association between high-risk HPV and anus neoplasm in men and women with immunodeficiency or immunosuppression has been confirmed and measures related to surveillance are standardized.

In patients without immunodeficiencies, this association is still unclear, which may contribute to the lack of adequate standards to diagnose HPV and prevent cancer of the anus.

The frequency of the cancer of anus previously considered low, is currently in considerable elevation, mainly squamous cell carcinoma (SCC).

The causal relationship between this virus and cancer of the cervix and the anus is established. These facts have motivated the inclusion of this disease as STD, which justifies the necessity of adopting surveillance measures in the clinics of sexual, gynecological and urological diseases.

Cancer of the anus, when diagnosed in the early stage, makes healing possible with less aggressive treatments, but in the advanced stage, abdominoperineal amputation is necessary.

Concerned about possible anal cancer, some gynecologists have referred patients with genital HPV to search for anal infection.

ELIGIBILITY:
Inclusion Criteria:

Female patients aged 18-65 years with an anatomic pathology compatible with CIN II / CIN III, without restriction regarding skin color, race, ethnicity, religion; Patients of the Oncology Gynecology Service of the HCSL, registered in the hospital management system, in outpatient consultations; Those who agree to participate in the study and sign the ICF. Patients attended at the general gynecological surgery outpatient clinic (control group) with no evidence of colpocitological alteration.

-

Exclusion Criteria:

Patients who withdraw the consent term. History of previous anal cancer / anal intraepithelial neoplasia. Immunosuppressed: HIV, SLE, users of immunosuppressive and transplanted drugs.

-

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2017-08-02 (Actual); Primary Completion 2018-04-30 (Estimated); Study Completion 2018-05-31 (Estimated)

PRIMARY OUTCOMES:
Study of Anal Cytologies in Patients With High Grade Cervical Intraepithelial Neoplasia (CIN II and III) | Six months
  Search for alterations in the anal cytology of patients with CIN 2-3 in conventional and liquid based anal citology

CONTACTS AND LOCATIONS:
Overall Officials: Daniela F Veiga, Study Chair — Vale do Sapucai University
Locations (1):
- Lyliana C R Barbosa, Pouso Alegre, Minas Gerais, Brazil

IPD SHARING:
Plan to Share IPD: No